CLINICAL TRIAL: NCT00095017
Title: A 4 Week Randomized, Placebo-Controlled, Parallel Group, Double-Blind Pilot Study to Assess the Safety and Efficacy of Etoricoxib 90 mg Versus Placebo in the Treatment of Cancer Pain
Brief Title: Safety and Efficacy of an Investigational Drug Versus Placebo in the Treatment of Cancer Pain (0663-083)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0663-083; 2004_090
Record Dates: First submitted 2004-10-29; First posted 2004-11-01 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Bone Neoplasms
Keywords: Arcoxia
MeSH Terms: conditions — Bone Neoplasms | interventions — Etoricoxib; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0663, etoricoxib / Duration of Treatment: 4 weeks

SUMMARY:
The purpose of this study is to compare the effectiveness of an investigational drug versus placebo in the treatment of metastatic bone cancer pain in patients diagnosed with breast or prostate cancer and a bone neoplasm. Patients in the study will be taking opioids to treat moderate to severe pain for their bone metastases and will remain on their opioids during the entire course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients are required to have a diagnosis of breast or prostate cancer with bone involvement and moderate to severe pain that requires opioid treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-11

PRIMARY OUTCOMES:
Analgesic efficacy over a 4 week treatment period; Safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC